CLINICAL TRIAL: NCT02722772
Title: Efficacy of Intra-Articular Injection of Etanercept for Moderate and Severe Knee Osteoarthritis
Acronym: EIAIETNKOA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Collaborators: Shanghai baiying pharmaceutical technology Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IAI-ETN-KOA-201613
Record Dates: First submitted 2016-03-24; First posted 2016-03-30 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-02

CONDITIONS: Osteoarthritis of Knee
Keywords: Intra-Articular Injection; Etanercept; TNF-α; IL-1; Osteoarthritis of Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Etanercept; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Etanercept treatment group (Experimental): Intra-articular injection of etanercept of 25 mg/w/joint and Health education, exercise and diet guidance; treatment: 5 weeks (If both knees are involved, the more significant symptomatic side is chosen for injection by etanercept)
  Interventions: Drug: Etanercept; Other: Health education, exercise and diet guidance
- Routine care group (Placebo Comparator): Health education, exercise and diet guidance; treatment: 5 weeks
  Interventions: Other: Health education, exercise and diet guidance

INTERVENTIONS:
Drug: Etanercept — Intra-articular injection of etanercept of 25mg/w/joint for 5 weeks.
  Arms: Etanercept treatment group
Other: Health education, exercise and diet guidance — Health education, exercise and diet guidance in patient; treatment: 5 weeks

SUMMARY:
Primary aim: evaluate efficacy of intra-articular injection of etanercept for moderate and severe knee osteoarthritis.

Second aim: investigate the potentiality of serum cytokines (TNF-α, Interleukin 1-α (IL1-α), IL1-β, matrix metalloproteinases1 (MMP1), MMP13) to predict the response of intra-articular injection of etanercept for moderate and severe knee osteoarthritis.

DETAILED DESCRIPTION:
1. Background:

   Osteoarthritis (osteoarthritis, OA) is a common joint disease. It is characterized by recurrent joint pain, swelling, increasing of disease status, joint deformity and activity disorders. [1]

   The pathogenesis of OA has not been fully understood. It may be associated with a variety of factors, such as: mechanics, biochemistry, genetics, and so on. Its main feature is the imbalance between synthesis and catabolism of articular cartilage cells. The imbalance may refer to cell aging, cell apoptosis, local inflammatory factor in joints as well as stress mechanism and so on. [2] OA usually develops in burdened and active joints, such as: the knee, the spine (cervical and lumbar spine), hip and ankle, hand joints, etc. The first session of The National Health and Nutrition Survey (The first National Health and Nutrition Examination Survey, NHANESI) found that 12% of people in The United States have at least one joint in accordance with the clinical diagnosis of OA. [3] Radiographic result shows that rate of American adults knee OA prevalence is 14% and 37%, and women are more common (4-6). A large study found that at least one joint in people over 55 years have radiographic hand OA, and female prevalence is 67%, male is 55% [7].

   The OA in Chinese are more likely happened in elder women than men. Prevalence rate could up to 50% in people over the age of 60, and 80% in 75 years old.

   Osteoarthritis patients suffer huge pain, and it cause huge economic burden to the society, and it becomes a serious impact on social productivity and lead to huge economic burden [8].

   In the United States, OA cost $ 1,855 billion per year and in 27 million patients, and women spend $ 6212 per year, male $ 4730 per year [2]; OA cost 1% ~ 2.5% of gross domestic product (GDP) in the United States, Britain, France, Canada, Australia and other developed countries. There is no burden of economic data of OA in China [9].

   Classification criteria of knee osteoarthritis

   According to the affected areas, OA can be divided into knee OA, hip OA, hand OA (distal interphalangeal joints, the first wrist palm joints), foot OA (first plantar toe joints, heel), etc.

   Knee OA is the most common disease in clinical disease. The classification of the knees OA contains clinical criteria, and also clinical and imaging criteria in the modified American College of Rheumatology (ACR) classification criteria in osteoarthritis classification criteria [10].

   Knee osteoarthritis usually occurs with obvious fricatives, bony enlargement, Baker cyst expansion and joint effusion is generally not associated with skin redness.

   The most common deformity comes out with varus in severe cases, but also it may appear in the early mild disease. That clinically obvious varus may be a predictive factor during the disease progression [11]. That quadriceps become weak is a changeable risk factor for early knees OA disease progression, especially in women (12-13). Muscle atrophy occurs in late stage of disease progression [14] [15]. And it brings huge burden of disease to patients.

   Treatment of knee OA

   The aim of the treatment is to relieve pain, prevent and delay the progress of disease, protect the joints function, improve the quality of life. The treatment should be individualized. Full consideration to the patient' illness risk factors should be given, including: joint structure changing, the degree of inflammation and pain, concurrent disease status and other specific situation and condition. Treatment should be given priority to combine non-drug therapy with drug therapy. Operation should be performed when it is necessary [16].

   Non-drug therapy include psychosocial intervention [16], decreasing weight [17], reasonable exercise [18], physical therapy which includes heat therapy, spa therapy, etc.), etc.

   Drug therapy mainly includes drugs using external, drugs using in whole body and drugs intra-articular injections [16].

   Topical drugs include: capsaicin [19], non-steroid anti-inflammatory drugs (NSAIDS) for external use [20] and lidocaine for external use only.

   Systemic medicine include: a: non-opiate drug. Acetaminophen is the first choice of OA treatment, and the main reason is that the less side effects and good curative effect [21].b: NSAIDS. There are two effect of NSAIDS: anti-pain and anti-inflammatory, which is the most commonly used for the control of OA symptoms. The main adverse reactions are gastrointestinal symptoms, renal or liver damage, effect on platelet function, and it may increase the risk of cardiovascular adverse events [22]. c: opioid analgesics. It can be considered if Pain still difficult to control after non-drug and drug treatment.

   Drugs injection intra-articular, including: intra-articular injection of glucocorticoid and hyaluronic acid derivatives [23].

   Research of TNF-α application in OA:

   TNF-α and IL1 play an important role in the pathogenesis of osteoarthritis, IL1 - beta often express highly in middle to late course of OA [24 to 27]. In the OA flare course, TNF-α and IL1 alpha will increase significantly; TNF-α has been considered to be one of the important factors associated with the degree of OA inflammatory, and the IL1 alpha has a significant relation with the start of OA inflammatory [27].
2. Aims:

   Primary: evaluate efficacy of intra-articular injection of etanercept for moderate and severe knee osteoarthritis Second: investigate the potentiality of serum cytokines (TNF-α, L1-α, IL1-β, MMP1, MMP13) to predict the response of intra-articular injection of etanercept for moderate and severe knee osteoarthritis.
3. Patients:

   Recruit Patients of moderate and severe knee osteoarthritis, totally 60 patients (According with classification of "Clinical Image" of 1986 American college of rheumatology criteria in osteoarthritis of the knee )
4. Study Design:

   A 12-week, multi-center, open-labeled, randomized study. Moderately and severe knee osteoarthritis patients, total 60 patients (consider expulsion rate 15%)(According with classification of "Clinical Image" of 1986 American college of rheumatology criteria in osteoarthritis of the knee )

   The 60 patients will be randomly assigned into two groups:

   Etanercept treatment group: Intra-articular injection of etanercept of 25mg/w/joint and health education, exercise and diet guidance; treatment: 5 weeks Routine care group: Health education, exercise and diet guidance; treatment: 5 weeks (If both knees are involved, the more significant symptomatic side is chosen for injection by etanercept)

   This study has two stages:
   1. Screening/baseline period: - 4 weeks ~ 0 weeks;

      Patients should have signed informed consent form (ICF) before participating the study

      Obtain the history before treatment, medical records, disease history and demographic information of patients. And also perform pregnancy test (optional), HIV testing (optional), hepatitis B virus (HBV) detection (optional), hepatitis C virus (HCV) detection (optional), electrocardiogram examination, chest radiograph, tuberculin test (PPD) test, vital signs, physical examination, blood routine, urine routine and blood biochemical examination, imaging examination (anteroposterior/lateral of X-ray in knee joint, horizontal position/lateral projection/side lateral projection of ultrasound in knee, supine position in knee joint of MRI (optional, sagittal and coronary are commonly used), measure the erythrocyte sedimentation rate (ESR) and C reactive protein (CRP) and store serum in - 80 ℃ to detect serum protein markers level during baseline period, at the same time, keep the plasma to - 80 ℃.(refer to "9.3 lab operation"). Collect disease assessment result in baseline, and record the Visual Analog Pain Scale (VAS) pain score, MOS 12-item Short Form Health Survey (SF12) score, the knee injury and osteoarthritis score (KOOS score), 30 s - Chair Stand Test (CST) score, 40 m Fast-paced Walk Test (FPWT) score, ultrasonic relative index score and MRI relative index score.
   2. Follow-up:baseline to 12 weeks, during this period, two groups of participants will be treated with Intra-articular injection of etanercept of 25 mg/w/joint, health education, exercise and diet guidance or just health education, exercise and diet guidance separately. During this period 4 times follow-up will be performed at 2nd, 4th, 8th, 12th week.

   At 2nd week, vital signs will be recorded, pain VAS score, SF12 score, KOOS score, condition of drug combination and adverse events will be recorded.

   At 4th week, vital signs will be recorded, and blood routine, urine routine, blood biochemical, the ESR and CRP will be examined and recorded, imaging examination (horizontal position/lateral projection/side lateral projection of ultrasound in knee), and collect basic evaluation results such as: pain VAS score, SF12 score, KOOS score, 30 s - CST score, 40 m FPWT score, ultrasonic relative index score and condition of drug combination and adverse events will be recorded.

   At 8th week, 12th week, vital signs, blood routine, urine routine and blood biochemical will be examined and recorded and imaging examination will be performed (horizontal position/lateral projection/side lateral projection of ultrasound in knee or supine position of MRI in knee joint, (optional, and sagittal and coronary will be used as usual)). Measure the ESR and CRP and store serum in - 80 ℃ to detect serum protein markers level during baseline to 8th week and 12th week, at the same time, store plasma to - 80 ℃.(refer to "9.3 lab operation"). Collect disease assessment result, and record the pain VAS score, SF12 score, KOOS score, 30 s - CST score, 40 m FPWT score, ultrasonic index score and MRI relative index score (optional). And condition of drug combination and adverse events will be recorded.
5. Laboratory tests

   Main laboratory examination:

   Detect the level of TNF-α, L1-α, IL1-β, MMP1, MMP13 levels in patients peripheral blood at baseline period and 4th week, 8th week by using enzyme-linked immunosorbent assay.
6. The curative effect evaluation/check points:

   The primary checkpoint: at 8th week and 12th week, changes of pain VAS score, KOOS score relative to the baseline.

   The Secondary checkpoints: at 8 weeks and 12 weeks changes of SF12 score, 30s-CST score, 40 m FPWT score, ultrasound score, MRI score, level of TNF alpha, IL1 alpha, IL1 - beta, MMP1, MMP13 in serum relative to the baseline.
7. Statistical methods:

Based on the curative effect data of patients, analysis by using R software or Statistical Analysis System (SAS) statistical software:

Calculate the measurement data using t-test and rank test; and rate is calculated using chi-square test.

Perform single factor and multiple factors regression analysis on indicators of baseline prognostic factors of patients (protein markers) and curative effect.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give full consent;
2. According with classification of "Clinical Image" of 1986 American college of rheumatology criteria in osteoarthritis of the knee ;
3. Grade II-III of Kellgren-Lawrence (KL) grading system, revealing synovial inflammation or synovial fluid by combining ultrasound and/or MRI
4. Knee pain for at least 1 Month and Pain VAS Score>4 during the last week;
5. Fertile women agreed to adopt effective contraceptive measures during the test.

Exclusion Criteria:

1. Allergic to pharmaceutical ingredients;
2. Received Tumor Necrosis Factor inhibitor (TNFI) or other biologics preparation within 3 months;
3. Received physical therapy or articular injection, taking antidepressants or antispasmodic, opioids within 3 months ;
4. Patients with history of knee surgery or upcoming surgery within 10 years;
5. Patients accompanied by other complications or joint disease (such as septic arthritis, osteonecrosis,haemochromatosis, ochronosis, etc.);
6. Patients with serious joint deformation or joint deformities;
7. Patients with active or a history of recurrent infections;
8. Patients existing active tuberculosis (TB) or has a history of active TB;
9. Patients with positive on hepatitis b surface antigen or hepatitis c antibody;
10. Patients with a history of severe lung disease, tumor;
11. Patients with severely abnormal function on liver and kidney (liver enzyme > = 2 times normal, creatinine > = normal);
12. Patients with pregnancy, ready for pregnancy or lactation;
13. Patients with other conditions which not suitable for use of Etanercept.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-07 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Pain VAS score(Pain Visual Analogue Scale/Score) | baseline to 8 weeks and 12 weeks
  Changes from the baseline to 8 weeks and 12 weeks to evaluate the treatment efficacy
KOOS score(The Knee injury and Osteoarthritis Score) | baseline to 8 weeks and 12 weeks
  Changes from the baseline to 8 weeks and 12 weeks to evaluate the treatment efficacy

SECONDARY OUTCOMES:
30s-CST score(30 seconds Sit/chair Test) | baseline to 8 weeks and 12 weeks
  Changes from the baseline to 8 weeks and 12 weeks to evaluate the activity of knee joint
40m FPWT score(40 meters fast walking test) | baseline to 8 weeks and 12 weeks
  Changes from the baseline to 8 weeks and 12 weeks to evaluate the activity of knee joint
Assessment score under ultrasound | baseline to 8 weeks and 12 weeks
  Changes from the baseline to 8 weeks and 12 weeks to evaluate the changes of patients' inner-structure of knee
Assessment score under MRI | baseline to 8 weeks and 12 weeks
  Changes from the baseline to 8 weeks and 12 weeks to evaluate the changes of patients' inner-structure of knee
TNF-α (pg/ml) level in serum | baseline to 8 weeks and 12 weeks
  Changes from the baseline to 8 weeks and 12 weeks to evaluate patients' inflammatory level
IL1-α (pg/ml) level in serum | baseline to 8 weeks and 12 weeks
  Changes from the baseline to 8 weeks and 12 weeks to evaluate patients' inflammatory level
IL1-β (pg/ml) level in serum | baseline to 8 weeks and 12 weeks
  Changes from the baseline to 8 weeks and 12 weeks to evaluate patients' inflammatory level
MMP1 (ng/ml) level in serum | baseline to 8 weeks and 12 weeks
  Changes from the baseline to 8 weeks and 12 weeks to evaluate patients' inflammatory level
MMP13 (ng/ml) level in serum | baseline to 8 weeks and 12 weeks
  Changes from the baseline to 8 weeks and 12 weeks to evaluate patients' inflammatory level
SF-12 score(MOS 12-item Short Form Health Survey) | baseline to 8 weeks and 12 weeks
  Changes from the baseline to 8 weeks and 12 weeks to evaluate patients' health condition

OTHER OUTCOMES:
Adverse event | 2 weeks, 4 weeks, 8 weeks and 12 weeks
  Type and frequency of adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyi Zhang, Study Chair — First Affiliated Hospital of Harbin Medical University; Yifang Mei, M.D, Principal Investigator — First Affiliated Hospital of Harbin Medical University
Locations (1):
- The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have not yet decided whether to share participants' data or not.

REFERENCES:
- [Background] Ge Z, Hu Y, Heng BC, Yang Z, Ouyang H, Lee EH, Cao T. Osteoarthritis and therapy. Arthritis Rheum. 2006 Jun 15;55(3):493-500. doi: 10.1002/art.21994. No abstract available. PMID 16739189
- [Background] Loeser RF, Goldring SR, Scanzello CR, Goldring MB. Osteoarthritis: a disease of the joint as an organ. Arthritis Rheum. 2012 Jun;64(6):1697-707. doi: 10.1002/art.34453. Epub 2012 Mar 5. No abstract available. PMID 22392533
- [Background] Lawrence RC, Felson DT, Helmick CG, Arnold LM, Choi H, Deyo RA, Gabriel S, Hirsch R, Hochberg MC, Hunder GG, Jordan JM, Katz JN, Kremers HM, Wolfe F; National Arthritis Data Workgroup. Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. Part II. Arthritis Rheum. 2008 Jan;58(1):26-35. doi: 10.1002/art.23176. PMID 18163497
- [Background] Dillon CF, Rasch EK, Gu Q, Hirsch R. Prevalence of knee osteoarthritis in the United States: arthritis data from the Third National Health and Nutrition Examination Survey 1991-94. J Rheumatol. 2006 Nov;33(11):2271-9. Epub 2006 Oct 1. PMID 17013996
- [Background] Felson DT, Naimark A, Anderson J, Kazis L, Castelli W, Meenan RF. The prevalence of knee osteoarthritis in the elderly. The Framingham Osteoarthritis Study. Arthritis Rheum. 1987 Aug;30(8):914-8. doi: 10.1002/art.1780300811. PMID 3632732
- [Background] Jordan JM, Helmick CG, Renner JB, Luta G, Dragomir AD, Woodard J, Fang F, Schwartz TA, Abbate LM, Callahan LF, Kalsbeek WD, Hochberg MC. Prevalence of knee symptoms and radiographic and symptomatic knee osteoarthritis in African Americans and Caucasians: the Johnston County Osteoarthritis Project. J Rheumatol. 2007 Jan;34(1):172-80. PMID 17216685
- [Background] Dahaghin S, Bierma-Zeinstra SM, Ginai AZ, Pols HA, Hazes JM, Koes BW. Prevalence and pattern of radiographic hand osteoarthritis and association with pain and disability (the Rotterdam study). Ann Rheum Dis. 2005 May;64(5):682-7. doi: 10.1136/ard.2004.023564. Epub 2004 Sep 16. PMID 15374852
- [Background] McCarberg B, Tenzer P. Complexities in the pharmacologic management of osteoarthritis pain. Curr Med Res Opin. 2013 May;29(5):539-48. doi: 10.1185/03007995.2013.785391. Epub 2013 Apr 3. PMID 23489409
- [Background] Kotlarz H, Gunnarsson CL, Fang H, Rizzo JA. Insurer and out-of-pocket costs of osteoarthritis in the US: evidence from national survey data. Arthritis Rheum. 2009 Dec;60(12):3546-53. doi: 10.1002/art.24984. PMID 19950287
- [Background] Altman R, Asch E, Bloch D, Bole G, Borenstein D, Brandt K, Christy W, Cooke TD, Greenwald R, Hochberg M, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. Arthritis Rheum. 1986 Aug;29(8):1039-49. doi: 10.1002/art.1780290816. PMID 3741515
- [Background] Chang A, Hochberg M, Song J, Dunlop D, Chmiel JS, Nevitt M, Hayes K, Eaton C, Bathon J, Jackson R, Kwoh CK, Sharma L. Frequency of varus and valgus thrust and factors associated with thrust presence in persons with or at higher risk of developing knee osteoarthritis. Arthritis Rheum. 2010 May;62(5):1403-11. doi: 10.1002/art.27377. PMID 20213800
- [Background] Segal NA, Glass NA, Torner J, Yang M, Felson DT, Sharma L, Nevitt M, Lewis CE. Quadriceps weakness predicts risk for knee joint space narrowing in women in the MOST cohort. Osteoarthritis Cartilage. 2010 Jun;18(6):769-75. doi: 10.1016/j.joca.2010.02.002. Epub 2010 Feb 11. PMID 20188686
- [Background] Baker KR, Xu L, Zhang Y, Nevitt M, Niu J, Aliabadi P, Yu W, Felson D. Quadriceps weakness and its relationship to tibiofemoral and patellofemoral knee osteoarthritis in Chinese: the Beijing osteoarthritis study. Arthritis Rheum. 2004 Jun;50(6):1815-21. doi: 10.1002/art.20261. PMID 15188358
- [Background] Slemenda C, Brandt KD, Heilman DK, Mazzuca S, Braunstein EM, Katz BP, Wolinsky FD. Quadriceps weakness and osteoarthritis of the knee. Ann Intern Med. 1997 Jul 15;127(2):97-104. doi: 10.7326/0003-4819-127-2-199707150-00001. PMID 9230035
- [Background] Ikeda S, Tsumura H, Torisu T. Age-related quadriceps-dominant muscle atrophy and incident radiographic knee osteoarthritis. J Orthop Sci. 2005;10(2):121-6. doi: 10.1007/s00776-004-0876-2. PMID 15815857
- [Background] Messier SP, Loeser RF, Mitchell MN, Valle G, Morgan TP, Rejeski WJ, Ettinger WH. Exercise and weight loss in obese older adults with knee osteoarthritis: a preliminary study. J Am Geriatr Soc. 2000 Sep;48(9):1062-72. doi: 10.1111/j.1532-5415.2000.tb04781.x. PMID 10983905
- [Background] Topp R, Woolley S, Hornyak J 3rd, Khuder S, Kahaleh B. The effect of dynamic versus isometric resistance training on pain and functioning among adults with osteoarthritis of the knee. Arch Phys Med Rehabil. 2002 Sep;83(9):1187-95. doi: 10.1053/apmr.2002.33988. PMID 12235596
- [Background] McCarthy GM, McCarty DJ. Effect of topical capsaicin in the therapy of painful osteoarthritis of the hands. J Rheumatol. 1992 Apr;19(4):604-7. PMID 1375648
- [Background] Dreiser RL, Tisne-Camus M. DHEP plasters as a topical treatment of knee osteoarthritis--a double-blind placebo-controlled study. Drugs Exp Clin Res. 1993;19(3):117-23. PMID 8112200
- [Background] Bradley JD, Brandt KD, Katz BP, Kalasinski LA, Ryan SI. Comparison of an antiinflammatory dose of ibuprofen, an analgesic dose of ibuprofen, and acetaminophen in the treatment of patients with osteoarthritis of the knee. N Engl J Med. 1991 Jul 11;325(2):87-91. doi: 10.1056/NEJM199107113250203. PMID 2052056
- [Background] Solomon SD, McMurray JJ, Pfeffer MA, Wittes J, Fowler R, Finn P, Anderson WF, Zauber A, Hawk E, Bertagnolli M; Adenoma Prevention with Celecoxib (APC) Study Investigators. Cardiovascular risk associated with celecoxib in a clinical trial for colorectal adenoma prevention. N Engl J Med. 2005 Mar 17;352(11):1071-80. doi: 10.1056/NEJMoa050405. Epub 2005 Feb 15. PMID 15713944
- [Background] Petrella RJ, DiSilvestro MD, Hildebrand C. Effects of hyaluronate sodium on pain and physical functioning in osteoarthritis of the knee: a randomized, double-blind, placebo-controlled clinical trial. Arch Intern Med. 2002 Feb 11;162(3):292-8. doi: 10.1001/archinte.162.3.292. PMID 11822921
- [Background] Goldring MB. The role of the chondrocyte in osteoarthritis. Arthritis Rheum. 2000 Sep;43(9):1916-26. doi: 10.1002/1529-0131(200009)43:93.0.CO;2-I. No abstract available. PMID 11014341
- [Background] Hunter DJ, Felson DT. Osteoarthritis. BMJ. 2006 Mar 18;332(7542):639-42. doi: 10.1136/bmj.332.7542.639. No abstract available. PMID 16543327
- [Background] Rai MF, Rachakonda PS, Manning K, Vorwerk B, Brunnberg L, Kohn B, Schmidt MF. Quantification of cytokines and inflammatory mediators in a three-dimensional model of inflammatory arthritis. Cytokine. 2008 Apr;42(1):8-17. doi: 10.1016/j.cyto.2008.02.004. Epub 2008 Mar 17. PMID 18343681
- [Background] Towle CA, Hung HH, Bonassar LJ, Treadwell BV, Mangham DC. Detection of interleukin-1 in the cartilage of patients with osteoarthritis: a possible autocrine/paracrine role in pathogenesis. Osteoarthritis Cartilage. 1997 Sep;5(5):293-300. doi: 10.1016/s1063-4584(97)80008-8. PMID 9497936